CLINICAL TRIAL: NCT06474091
Title: Liquid Biopsy MonitORing Of CholangioCarcinOma for Treatment Response and Prognostic Outcomes (MOROCCO)
Status: Enrolling by invitation | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 23-013283; NCI-2024-04798 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 23-013283 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2024-06-19; First posted 2024-06-25 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Cholangiocarcinoma
MeSH Terms: conditions — Cholangiocarcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples retained with permission of participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational: Patients undergo collection of blood samples and have their medical records reviewed on study. Patients also undergo collection of archived tissue samples on study.
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — Non-Interventional Study

SUMMARY:
This study explores the potential value of a new blood test approach to detect measurable residual disease or early recurrence/progression in patients with cholangiocarcinoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the association of PUMA levels from peripheral blood with disease progression (radiographically or clinically) in patients that are candidates for curative surgical intervention of cholangiocarcinoma.

Ia. Pre- and post-neoadjuvant-treatment PUMA levels will be associated with treatment response to neoadjuvant therapy (short term progression).

Ib. Pre-surgical and post-surgical PUMA levels will be associated with progression free survival.

II. To estimate the association of PUMA levels from peripheral blood with postoperative survival in patients treated for cholangiocarcinoma.

OUTLINE: This is an observational study.

Patients undergo collection of blood samples and have their medical records reviewed on study. Patients also undergo collection of archived tissue samples on study.

ELIGIBILITY:
Inclusion Criteria:

* Patient has a suspected or clinical diagnosis cholangiocarcinoma and under evaluation for surgical intervention with intent to cure
* Age ≥ 18 years

Exclusion Criteria:

* Patient has metastatic disease involving other organs (excluding lymph node)
* Patent has known primary cancer outside of the bile ducts within the last 3 years prior to blood collection (not including basal cell or squamous cell skin cancers, indolent cancer not requiring treatment within 3 years i.e. kidney, prostate or thyroid being observed)
* Patient has had surgery to remove current target pathology completely or partially
* Patient has undergone any prior radiation therapy to target lesion prior to blood collection
* Patient has received chemotherapy class drugs in the 3 years prior to blood collection
* Patient has had any transplants prior to blood collection
* Current target pathology is a recurrence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a clinical diagnosis of cholangiocarcinoma under evaluation for surgical intervention with intent to cure.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-05-08 (Actual); Primary Completion 2029-05-08 (Estimated); Study Completion 2029-05-08 (Estimated)

PRIMARY OUTCOMES:
Associate of PUMA levels with short term progression | Up to 5 years
  Proteins, mUtations, Methylated DNA, and Aneuploidy (PUMA) markers will be assessed pre- and post-treatment and will be associated with treatment response to therapy (short term progression; time to cholangiocarcinoma recurrence).
Associate of PUMA levels with progression free survival | Up to 5 years
  Pre-surgical and post-surgical PUMA levels will be associated with progression free survival (time to death from cholangiocarcinoma).

CONTACTS AND LOCATIONS:
Overall Officials: Nguyen H. Tran, MD, Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials